CLINICAL TRIAL: NCT05833893
Title: Clinical Study of XPO1 Inhibitor Selinexor Combined With COPL in Newly Diagnosed Advanced NK/T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhao, Chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XCOPL - NK/T -P01
Record Dates: First submitted 2023-02-25; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: nk/T-cell Lymphoma; Newly Diagnosed; Advanced Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): COPL + XPO1 inhibitor (Selinexor, 60 mg, po., d1,8,15)
  Interventions: Drug: XPO1 inhibitor

INTERVENTIONS:
Drug: XPO1 inhibitor — COPL + XPO1 inhibitor (Selinexor, 60 mg, po., d1,8,15)
  Other Names: COPL

SUMMARY:
Patients with newly diagnosed, pathologically confirmed NK/T-cell lymphoma of stage III-IV treated with XCOPL regimen. 3 weeks for a cycle, with a total of 6-8 cycles.

DETAILED DESCRIPTION:
Patients with newly diagnosed, pathologically confirmed NK/T-cell lymphoma of stage III-IV treated with XCOPL regimen. 3 weeks for a cycle, with a total of 6-8 cycles. Initial safety and PET-CT assessment were performed after 3 cycles of treatment (which could be delayed until 4 cycles of treatment in special cases). Patients who achieved partial remission or above will continue the original regimen, and patients who did not achieve partial remission or above will perform re-biopsy and be excluded from the group. Patients who remain partial remission by PET-CT evaluation after 6 cycles may switch to a second-line regimen (referring to NCCN guidelines, GDP regimen combined with selinexor is recommended). Chemotherapy will be performed for up to 8 cycles (followed by autologous or allogeneic hematopoietic stem cell transplantation), after which follow-up period was entered. It is recommended to perform ultrasound or CT evaluation, peripheral blood ctDNA and EBV copy number every three months during the first year of follow-up, and PET-CT evaluation every half a year.

ELIGIBILITY:
Inclusion Criteria:

* Age≥14 years, male or female;
* Pathologically confirmed newly diagnosed NK/T cell lymphoma according to WHO classification criteria 2016;
* At least one measurable lesion, defined as bidimensionally measurable, intranodal lesion > 1.5 cm in short axis and extranodal lesion > 1.0 cm in short axis;
* ECOG score 0~2;
* Clinical stage III~IV;
* Normal major organ function, meeting the following definitions: Hematology: WBC ≥ 3.5 x 10 9/L, PLT ≥ 75 x 10 9/L, Hb ≥ 80 g/L; Liver and kidney function: AST and ALT ≤ 3.0 ULN; TBIL ≤ 2.0 mg/dL; CCr ≥ 60 mL/min; liver and kidney function impairment caused by tumor compression is not limited by this; Fibrinogen: normal at first cycle
* Expected survival > 6 months
* Agree to use effective contraception;
* Understand and voluntarily sign written informed consent

Exclusion Criteria:

* Prior allogeneic HCT (allo-HCT)
* Active autoimmune disease
* Primary central nervous system lymphoma;
* Patients with infection which requiring treatment. Could be re-enrollment after infection control;
* Known history of human immunodeficiency virus (HIV) infection
* Known hypersensitivity to the study drug or any of its excipients;
* Presence of other active malignancy requiring treatment that could interfere with this study;
* Patients with other conditions not suitable for enrollment as judged by the investigator.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
response rate | 1-year
  complete remission + partial remission
Incidence of Treatment-Emergent Adverse Events | 1-year
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
the 1-year PFS | 1-year
  To evaluate the 1-year PFS of XCOPL regimen in advanced NK/T-cell lymphoma
the 1-year OS | 1-year
  To evaluate the 1-year OS of XCOPL regimen in advanced NK/T-cell lymphoma
the ctDNA and EBV copy number in peripheral blood | 1-year
  To evaluate the feasibility of measurable residual disease (MRD) detection and clinical recurrence prediction by ctDNA and EBV copy number.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhao, Graduate, Principal Investigator — Chief; Sai Huang, Graduate, Principal Investigator — Attending doctor
Locations (1):
- ChinaPLAGH, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No
Clinical study of XPO1 inhibitor Selinexor combined with COPL in newly diagnosed advanced NK/T-cell lymphoma

REFERENCES:
- [Result] Benkova K, Mihalyova J, Hajek R, Jelinek T. Selinexor, selective inhibitor of nuclear export: Unselective bullet for blood cancers. Blood Rev. 2021 Mar;46:100758. doi: 10.1016/j.blre.2020.100758. Epub 2020 Sep 15. PMID 32972802
- [Result] Tse E, Kwong YL. Diagnosis and management of extranodal NK/T cell lymphoma nasal type. Expert Rev Hematol. 2016 Sep;9(9):861-71. doi: 10.1080/17474086.2016.1206465. Epub 2016 Jul 8. PMID 27347812
- [Result] Lim SH, Hong JY, Lim ST, Hong H, Arnoud J, Zhao W, Yoon DH, Tang T, Cho J, Park S, Ko YH, Kim SJ, Suh C, Lin T, Kim WS. Beyond first-line non-anthracycline-based chemotherapy for extranodal NK/T-cell lymphoma: clinical outcome and current perspectives on salvage therapy for patients after first relapse and progression of disease. Ann Oncol. 2017 Sep 1;28(9):2199-2205. doi: 10.1093/annonc/mdx316. PMID 28911074